CLINICAL TRIAL: NCT07011277
Title: Investigation of Gait Characteristics in Women With Breast Cancer Related Lymphedema
Brief Title: Gait Characteristics of Women With Breast Cancer-Related Lymphedema
Status: Enrolling by invitation | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ilke Keser, Professor, Physical Therapist, Gazi University
Other Study IDs: Breast Cancer-Gait Analysis
Record Dates: First submitted 2025-05-18; First posted 2025-06-08 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Related Lymphedema
Keywords: breast cancer; lymphedema; gait disorders; upper extremity disorders
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms; Lymphedema; Mobility Limitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Women with breast cancer-related lymphedema
- Control group: Healthy women

SUMMARY:
Upper extremity lymphedema is one of the most common problems associated with cancer treatments in breast cancer survivors. Lymphedema causes asymmetry, changes posture, decreases arm swing due to increased weight, and as a result, may affects the patients' gait. The aim of this study is to examine the gait parameters in women with breast cancer-related lymphedema. Women diagnosed with breast cancer who are referred to the Gazi University Health Sciences Faculty Physiotherapy and Rehabilitation Department Oncological Rehabilitation Unit to receive physiotherapy recommendations and healthy volunteers will be included in the study. The demographic and clinical characteristics of the individuals will be recorded. Body Mass Index (BMI) will be calculated. Then, presence of lymphedema and lymphedema severity will be evaluated by measuring the circumference of the arms with a tape measure. Active shoulder joint movements will be evaluated with goniometer, handgrip strength with K-Force hand dynamometer, spatiotemporal parameters of gait and pelvic symmetry will be evaluated using BTS G-Walk wearable motion analysis system. Women with breast cancer related lymphedema will be compared with healthy women in terms of relevant parameters of gait. In addition, the relationship between lymphedema severity, shoulder joint movement limitation and grip strength with gait parameters in women with breast cancer and lymphedema will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Having breast cancer related lymphedema
* Being between the ages of 25-70
* Completing cancer treatments

Exclusion Criteria:

* Having orthopedic, neurological or vision problems that may affect walking
* Being in the active treatment process (being in the acute phase after surgery, receiving chemotherapy or radiotherapy)

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was conducted at the Oncological Rehabilitation Unit in Gazi University. Women with breast cancer related lymphedema (study group) who were referred to receive physiotherapy recommendations were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Lymphedema Severity | baseline
  Lymphedema will be assessed by measuring the circumference according to Kuhnke's disc method. The circumference measurement will be assessed by starting from the styloid process of the ulna with a tape measure and extending to the axilla at 4 cm intervals. Lymphedema diagnosis will be confirmed by a difference of more than 2 cm between both extremities and will be classified as mild for differences between both extremities were less than 3 cm, moderate for 3-5 cm and severe for more than 5 cm
Shoulder Range of Motion | baseline
  The patients' active shoulder flexion, abduction, external rotation and internal rotation range of motion will be measured in the supine position with a goniometer and record in degrees.
Handgrip Strength | baseline
  Patients' handgrip strength will be assessed with the K-force Grip dynamometer (Kinvent, Montpellier, France). Patients will be positioned to sit with the shoulder adducted, the elbow flexed at 90°, and the forearm in a neutral position. A total of three measurements will be taken from each patient, and the average of the three measurements will be recorded in kg.
Spatio-temporal Gait Characteristics | baseline
  Gait will be assessed using the BTS G-Walk (BTS Bioengineering, Italy). For gait analysis, a wireless inter-sensor system will be placed at the level of the 5th lumbar vertebra with a semi-elastic belt. This inertial system consists of a triaxial accelerometer, a triaxial magnetometer, a triaxial gyroscope and a GPS receiver. All data are collected at a frequency of 100 Hz and transmitted to a computer via a Bluetooth 3.0 connection. A specific software (BTS G-Studio) allows the processing of the information and the calculation of spatiotemporal gait parameters.
Pelvic Symmetry in Gait | baseline
  Pelvic symmetry will be assed with BTS G-Walk (BTS Bioengineering, Italy). For gait analysis, a wireless inter-sensor system will be placed at the level of the 5th lumbar vertebra with a semi-elastic belt. This inertial system consists of a triaxial accelerometer, a triaxial magnetometer, a triaxial gyroscope and a GPS receiver. All data are collected at a frequency of 100 Hz and transmitted to a computer via a Bluetooth 3.0 connection. A specific software (BTS G-Studio) allows the the processing of the information and the calculation of the percentage of pelvic symmetry between both limbs.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Health Sciences, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No